CLINICAL TRIAL: NCT01463514
Title: Noninvasive Determination Of Cerebral Tissue Oxygenation And Cerebral Blood Flow With Near-Infrared Spectroscopy In Patients With Pulmonary Hypertension Undergoing Right Heart Catheterization
Brief Title: Noninvasive Determination of Cerebral Tissue Oxygenation in Pulmonary Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NIRS_Study_1
Record Dates: First submitted 2011-10-18; First posted 2011-11-02 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension,; NIRS,; Near-infrared spectroscopy,; cerebral tissue oxygenation,; cerebral blood flow
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- AIR (Experimental): Randomization sequences according to modified catheter protocol.
  1. AIR 2. Target Oxygen(88-90%) 3. 100% Oxygen 4. Nitric Oxygen
  Interventions: Procedure: Right heart catheterization; Procedure: Near-infrared spectroscopy
- NO (Experimental): Randomization sequences according to modified catheter protocol.
  1.Nitric Oxygen 2. AIR 3. Target Oxygen(88-90%) 4. 100% Oxygen
  Interventions: Procedure: Right heart catheterization; Procedure: Near-infrared spectroscopy
- Oxygen (Experimental): Randomization sequences according to modified catheter protocol.
  1. 100% Oxygen 2. NO 3. AIR 4. Target Oxygen (88-90%)
  Interventions: Procedure: Right heart catheterization; Procedure: Near-infrared spectroscopy
- Target Oxygen (Experimental): Randomization sequences according to modified catheter protocol.
  1. Target Oxygen (88-90%) 2. 100% Oxygen 3. NO 4. AIR
  Interventions: Procedure: Right heart catheterization; Procedure: Near-infrared spectroscopy

INTERVENTIONS:
Procedure: Right heart catheterization — Oxygenation and hemodynamic parameters will be assessed during RHC according to standard procedures. All measurements will be noted as usual for PH assessment including: at rest breathing room air, during an oxygen challenge, under vasodilator testing with NO and/or during exercise. Room air, supplemental oxygen and NO will be applied over common breathing mask while patient is in a supine position. Oxygen will be taken as usual from the common adjustable hospital wall access, NO will be taken according to usual clinical practice during RHC from a gas cylinder connected to a reservoir, where adequate ppm concentration can be regulated. A dose of 40 ppm NO will be used according to common practise. Oxygen delivery to maintain the peripheral oxygen saturation between 88% and 90% will be adjusted over a 3 minute period of time.
Procedure: Near-infrared spectroscopy — For study purpose, patients will have additional non-invasive NIRS assessment. The measurement will take place during right heart catheterization.
  Other Names: INVOS® device (SOMANETICS CORPORATION, TROY, MICHIGAN, USA

SUMMARY:
To study the effect of acute pulmonary vasodilatation on cerebral tissue oxygenation (CTO) and cerebral blood flow (CBF) as indicator for cerebrovascular autoregulation in comparison to the effects of supplemental oxygen, decreased carbon dioxide by hyperventilation and exercise in patients with pulmonary hypertension (PH) undergoing clinically indicated right heart catheterisation (RHC).

Oxygenation and hemodynamic parameters will be assessed during RHC according to standard procedures. Non-invasive near infrared spectroscopy (NIRS) and a nasal canula will be additionally applied to measure CTO, CBF and endtidal CO2 (EtCO2). All parameters will be obtained at rest breathing room air, during an oxygen challenge, during standardized hyperventilation, under vasodilatation testing and during exercise in random, single-blinded sequences (except for exercise and hyperventilation). Pulmonary, systemic and cerebral oxygenation parameters and hemodynamics will be correlated with each other and functional class, quality of life, exercise and cognitive assessments at the time of the RHC and after three month.

ELIGIBILITY:
Inclusion criteria: Inclusion criteria are age 18 years or older, to be scheduled for RHC due to suspected or known PH and the ability to give informed consent. Both genders will be accepted.

Exclusion criteria: Exclusion criteria are: inability to follow the study due to language or cognitive problems (e.g. a major active psychiatric disorders, prior traumatic brain injury, and neurologic disease), dementia on the basis of a Mini Mental State Test and pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Changes from baseline cerebral tissue oxygenation (in %) during right heart catheterization and after 3 month | First measurement (day 1 = day of examination) during right heart catherization and after 3 month (follow-up)
  Acute effects (deviation from baseline measurements in % of oxygenated blood) of oxygen challenge, hyperventilation and vasodilator testing during right heart catheterization on cerebral tissue oxygenation in patients with pulmonay hypertension
Changes in cerebral blood flow (in % from baseline) during right heart catheterization and after 3 month | First measurement (day 1 = day of examination) during right heart catherization and after 3 month (follow-up)
  Acute effects (deviation from baseline measurements in % from baseline) of oxygen challenge, hyperventilation and vasodilator testing during right heart catheterization on cerebral blood flow in patients with pulmonay hypertension

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich; Silvia Ulrich Somaini, MD, Principal Investigator — University Hospital Zurich, Division of Pneumology
Locations (1):
- University Hospital Zurich, Pneumology, Zurich, Switzerland

REFERENCES:
- [Derived] Muller-Mottet S, Hildenbrand FF, Keusch S, Hasler E, Maggiorini M, Speich R, Bloch KE, Ulrich S. Effects of exercise and vasodilators on cerebral tissue oxygenation in pulmonary hypertension. Lung. 2015 Feb;193(1):113-20. doi: 10.1007/s00408-014-9667-5. Epub 2014 Nov 21. PMID 25413133